CLINICAL TRIAL: NCT05589415
Title: Targeted High-Definition tDCS to Improve Upper Limb Rehabilitation in SCI
Brief Title: Targeted HD-tDCS to Improve Upper Limb Rehabilitation in SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-20-0326
Record Dates: First submitted 2022-06-23; First posted 2022-10-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Rehabilitation; Upper Limb; Brain Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Definition tDCS and rehabilitation (Experimental): 10 sessions (2 hours/session) will be completed with high definition tDCS and upper limb rehabilitation.
  Two times prior and two times after rehabilitation, upper limb weakness and neurophysiology will be assessed.
  Interventions: Device: High-definition Transcranial Direct Current Stimulation
- Conventional tDCS and rehabilitation (Active Comparator): 10 sessions (2 hours/session) will be completed with conventional tDCS and upper limb rehabilitation.
  Two times prior and two times after rehabilitation, upper limb weakness and neurophysiology will be assessed.
  Interventions: Device: Conventional Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High-definition Transcranial Direct Current Stimulation — High-definition Transcranial Direct Current Stimulation (HD-tDCS) delivers current through five small electrodes (0.8 cm2) placed in an "X-shaped" configuration via a simple cap. This configuration leads to an 80% greater concentration or focusing of the electric field within the targeted region compared to conventional, non-focal Transcranial Direct Current Stimulation (tDCS). The participant will undergo 30 minutes of treatment at 2 milliamps.
  Arms: High Definition tDCS and rehabilitation
Device: Conventional Transcranial Direct Current Stimulation — Surface electrodes will be placed in saline-soaked sponges (5 x 7 cm2) and applied to different regions of the scalp. The participant will undergo 30 minutes of treatment at 2 milliamps.
  Other Names: Transcranial Direct Current Stimulation
  Arms: Conventional tDCS and rehabilitation

SUMMARY:
The proposed project seeks to maximize the functional recovery achieved during the rehabilitation of the paretic upper limbs in individuals with SCI. The investigation will work towards optimizing the use of transcranial direct current stimulation (tDCS), an adjunct known to improve the effectiveness of rehabilitation. In particular, the relationship between the specificity of current delivery and functional benefit will be explored, and findings may lead to a framework that can be translated to the clinic setting.

DETAILED DESCRIPTION:
The investigators recently completed a clinical trial evaluating whether upper limb function in those with SCI could be improved by pairing rehabilitation with conventional tDCS. Overall, the investigators found that conventional tDCS showed promise in improving upper limb function, with an observed effect size ranging from 0.23 to 0.58. Using data from this trial, the investigators performed a retrospective analysis to determine whether the level of functional benefit the subject experienced was related to the strength of tDCS current delivered to the cortical areas dedicated to weak muscles. The investigators approximated the delivery of current using models from software developed by collaborator Dr. Bikson. The current investigators' analysis found that improvements in dexterity following ten sessions of conventional, non-focal (35 cm2) tDCS were greater when the current was delivered mainly within the motor cortical areas dedicated to the weak muscles.

Expanding on the retrospective analysis, the investigators have recently conducted a pilot study to determine whether focality of tDCS can directly change functional benefits in individuals with SCI. Specifically, the investigators conducted a single-session cross-over study evaluating the effect of conventional, sham, and a focused tDCS on grip strength and corticospinal pathway excitability (n=2). For the current study, the investigators utilized high-definition tDCS (HD-tDCS) to deliver a more focal current with tDCS. HD-tDCS delivers current through five small electrodes (0.8 cm2) placed in an "X-shaped" configuration via a simple cap. This configuration leads to an 80% greater concentration or focusing of the electric field within the targeted region compared to conventional, non-focal tDCS.

In the current cross-over study, outcomes were assessed before and immediately following a 30-minute application of tDCS paired with task training. Sessions were spaced one week apart to allow for sufficient wash-out. The Investigators found that HD-tDCS had a substantial impact on grip strength compared to conventional tDCS. Most notably, HD-tDCS improved grip strength (+15.9 N) while conventional tDCS reduced grip strength (-5.5 N). With the added grip strength following HD-tDCS, subjects reported the new ability to grip a bottle of water and hold small objects, indicating the greater potential for clinical impact compared to conventional tDCS. Overall, raw changes in grip strength translated to a 40% advantage of HD-tDCS compared to conventional tDCS, wherein a change greater than 15% was defined as clinically significant. The Investigators also observed that the single application of HD-tDCS could result in greater increases in corticospinal excitability of the weak triceps muscle compared to conventional tDCS. This is not surprising since focusing the electric field has been shown to elicit greater, longer-lasting increases in corticospinal excitability in healthy individuals; an effect that likely occurs since more current flow is less variable and arrives at cortical targets after HD-tDCS (98% improvement over conventional tDCS). Based on the investigators' previous findings, HD-tDCS is expected to deliver upwards of a 40% advantage and provide clinically significant gains compared to conventional tDCS for the proposed clinical trial.

The investigators' collective finding that focality of tDCS can directly change functional benefit and corticospinal excitability is corroborated by others. Of note, work in stroke aphasia has shown that targeting tDCS current to the cortical regions activated during speech improves the functional benefit of tDCS. Similar findings have been reported in fibromyalgia and working memory. Thus, in combination with others, the investigators' result provides the impetus to study whether the application of focal tDCS would lead to even greater improvements in upper limb function than that achieved with conventional, non-focal tDCS.

The current study will directly build off the investigators' initial clinical trial and pilot cross-over study. The investigators will perform a clinical feasibility trial and test for the first time whether the application of HD-tDCS in SCI elicits more robust increases in the excitability of residual corticospinal pathways and function of the paretic upper limbs than the application of conventional tDCS.

Twenty-four subjects with a chronic C2-C6 SCI will be enrolled in a randomized, assessor-blinded, clinical feasibility trial (See Section 1.3). Prior to randomization, subjects will complete a two-week baseline control phase. The data from the baseline control phase will allow each patient to serve as their own control since variability due to disease heterogeneity and tDCS can be accounted for in the data analysis. After completion of the baseline control phase, subjects will be randomized into two groups: HD-tDCS + massed practice training or conventional tDCS + massed practice training. Randomization will be performed using a generalized randomized block design. Subjects within a block will be matched on strength of the weak triceps (i.e., maximum volitional contraction measured by electromyography; EMG). Computer-based software for randomization will be used. Immediately after the intervention, subjects will undergo functional and neurophysiologic testing at post-test and follow-up (four weeks after intervention). Since conventional and HD-tDCS applications visually look different, only assessors collecting and analyzing the neurophysiologic and upper limb functional outcomes will be blinded to the tDCS paradigm delivered.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age between 18 and 75 years
* Physician diagnosed cervical incomplete spinal cord injury or lesion (iSCI)
* Classified by the American Spinal Cord Association (AIS) impairment scale as AIS C or D
* iSCI occurred at least 18 months ago
* Level of injury or lesion is between C2 and T1
* Bicep strength must be classified as ≥ 3 muscle grade as defined by the medical research council (MRC) scale
* Tricep strength must be at least an MRC grade of 2 and be at least 1 muscle grade lower than bicep
* Both the biceps and triceps will be required to elicit an active motor evoked potential >200 uV with transcranial magnetic stimulation
* Must maintain current medication regime
* Must present with a weaker side of the body, as indicated by a Upper Extremity Motor Score (UEMS) score difference between the left and right side
* UEMS < 40 (50 max score)

Exclusion Criteria:

* Pacemaker or other implanted device
* Metal in the skull
* History of seizures
* Pregnancy
* First-degree relative with medication-resistant epilepsy
* Current participation in upper limb rehabilitation therapies
* Current use of illicit drugs, abusing alcohol, or have withdrawn from alcohol in the last 6 months
* Other neurological impairment or condition
* Pressure ulcers
* Significant lower motor neuron loss at C7 as noted by a nerve conduction velocity <50 m/s
* History of traumatic brain injury, as documented by Rancho Scale Impairment of ≤ 5
* History of brain MRI documented focal cerebral cortex infarct (e.g. hydrocephalus)
* Contractures at the elbow
* Severe spasticity as noted by a Modified Ashworth Scale (MAS) > 4.
* Documented, non-sedated post-traumatic amnesia lasting more than 48 hours
* Demonstrated present gains in motor recovery as noted by a >10% change in triceps strength from pre-test #1 to pre-test #2
* A neuroactive medication that has the potential to lower the seizure threshold

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) | Collected four times during study duration: (Baseline-phase) Day 1 and 14; (Post-Rehabilitation-phase) Day 1 and 14
  Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) is a clinical tool that incorporates assessment of both upper limb motor function and activity limitations (9 hole peg test, grasping). The Investigators will assess the changes in movement control from Baseline, 2 weeks, and after four weeks of rehabilitation. An increase in time spent completing the peg test and grasping test signifies an increase in a participant's performance of strength, sensibility, and prehension.
Excitability of weak muscle pathways | Collected four times during study duration: (Baseline-phase) Day 1 and 14; (Post-Rehabilitation-phase) Day 1 and 14
  Using Transcranial Magnetic Stimulation (TMS) to promote Motor Evoked Potentials (MEP), the Investigators will monitor changes in cortical excitability of the weak muscle (Abductor Digiti Minimi; ADM) motor hotspot by measuring the muscle excitability with Electromyography (EMG; in millivolts) from Baseline, 2 weeks, and after four weeks of rehabilitation.
  The motor hotspot of the weak muscle will be defined as the site that evokes MEPs ≥50 mV at the lowest intensity (% device output), or the resting motor threshold (RMT). A decrease of the TMS's percentage output to promote MEPs of the weak muscle signifies a decrease in the cortical excitability, as measured by Active Motor Thresholds (AMT) and Active Motor Evoked Potentials (AMEP).

SECONDARY OUTCOMES:
Electromyography (EMG) Tracking Accuracy | Collected four times during study duration: (Baseline-phase) Day 1 and 14; (Post-Rehabilitation-phase) Day 1 and 14
  For the current task, subjects will be asked to match their weak muscle (Abductor Digiti Minimi; ADM) Electromyography (EMG) force to a sine wave with a peak and valley within their strength range displayed on a computer monitor. The investigators will then assess the changes in the subjects' accuracy of matching their EMG force to a sine wave from Baseline, 2-weeks, and after four weeks of rehabilitation. An increase in the variability of a participant keeping their weak muscle EMG force represented as a sine wave within the zone indicates a decrease in performance.
Maximum Volitional Contraction (MVC) | Collected four times during study duration: (Baseline-phase) Day 1 and 14; (Post-Rehabilitation-phase) Day 1 and 14
  The subjects will be asked to do a maximum contraction of their biceps followed by their triceps, and the investigators will assess the changes in their Maximum Volitional Contraction (MVC; in three trials) using Electromyography (EMG; Root Mean Square in millivolts) from Baseline, 2 weeks, and after four weeks of rehabilitation. A greater number of Root Mean Square millivoltage registered on the EMG signifies a higher MVC.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Baker, PhD, Principal Investigator — University of Texas Rio Grande Valley
Locations (1):
- University of Texas Rio Grande Valley, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data may be shared with interested researchers upon request. There is not a formal sharing plan in place.